CLINICAL TRIAL: NCT06048744
Title: Ultrasound Guided Erector Spinae Plane Block vs External Oblique Intercostal Plane Block for Postoperative Analgesia in Patients Undergoing Subcoastal Nephrectomy: A Randomised Trial
Brief Title: Ultrasound Guided Erector Spinae Plane Block vs External Oblique Intercostal Plane Block for Nephrectomy
Acronym: EOINBvsESB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9/2023ANET1-2
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- external oblique intercostal block (Active Comparator): After induction of general anesthesia, external oblique intercostal blocks will be performed with patients positioned in the supine position with their ipsilateral arm abducted.
  A 14-15 MHz linear ultrasound transducer (Sono-Site) was placed in the sagittal plane between the midclavicular and anterior axillary lines at the level of sixth rib.
  30 ml of bupivacaine 0.25% will be administered incrementally. The drug will be injected after a negative aspiration into the plane deep to the external oblique muscle and superficial to the sixth and seventh ribs and their associated intercostal muscles.
  Interventions: Procedure: external oblique intercostal block
- Erector Spine Block (Active Comparator): After induction of general anesthesia, patients will be positioned in the lateral position . A linear ultrasound transducer will be placed on the midline to identify the T8 spinous process. From this position, the ultrasound transducer was moved 2-3 cm laterally to visualize the hyperechoic line of the T8 transverse process with its associated acoustic shadow inferiorly, and the overlying erector spinae muscle superiorly. 30 ml 0.25% bupivacaine will be injected.
  Interventions: Procedure: Erector Spine block

INTERVENTIONS:
Procedure: external oblique intercostal block — U S guided external oblique intercostal block after induction.
  Arms: external oblique intercostal block
Procedure: Erector Spine block — US guided erector spine block after induction
  Arms: Erector Spine Block

SUMMARY:
The patients will be randomly allocated into two equal groups using a computer program.

Group A: will receive U S guided external oblique intercostal block after induction.

Group B:

Patients will receive US guided erector spine block after induction.

DETAILED DESCRIPTION:
Patients will be premedicated with IV midazolam (0.05 mg/kg). Under standard monitoring including Electrocardiography, Non-Invasive Blood Pressure, and Pulse Oximetry. General Anesthesia will be induced with Fentanyl (1-2 μg/kg), Propofol (2-3 mg/kg), and Atracurium (0.5-0.8 mg/kg). Pressure controlled Volume guarantee Ventilation mode will be used to maintain O2 Saturation Above 98%. Anesthesia will be maintained with Isoflurane 1.2 Minimum Alveolar Concentration inhalation

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be older than 21 years old with American society of anesthesiology ASA physical status I& II&III scheduled for elective (Subcostal) Nephrectomy

Exclusion Criteria:

* Patients who are:
* Uncooperative.
* Having allergy to any of the study drugs.
* Known abuse of alcohol or medication.
* Having Local infection at the site of injection or systemic infection.
* Pregnancy.
* With coagulation disorders or on anticoagulation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
time for first rescue analgesia | day 0
  hours

SECONDARY OUTCOMES:
visual analogue score VAS score | 24 hours
  (a scale from 0 to 10 where 0 is interpreted as no pain, 1-4 mild pain, 5-6 moderate pain, 7-10 severe pain) will be recorded 15 min after extubation (as soon as the patient will be alert enough to report pain)
the number of rescue analgesics | 24hours
  numbers'

CONTACTS AND LOCATIONS:
Overall Officials: AMAL G SAFAN, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: No